CLINICAL TRIAL: NCT02467504
Title: A Randomized, Double Blind, Placebo-controlled Pilot-study to Evaluate Efficacy and Safety of Low-dose hrIL-2 in the Treatment of Methotrexate (MTX)-Naive Patients With Rheumatoid Arthritis
Brief Title: Low-dose Recombinant Human IL-2 for the Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Monash University (Other); Beijing ShuangLu Pharmaceutical Co., Ltd. (Other)
Responsible Party: Principal Investigator, Zhanguo Li, Dept. Rheumatology and immunology,Peking University People's Hospital, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: hrIL-2 RA
Record Dates: First submitted 2015-06-04; First posted 2015-06-10 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Folic Acid; loxoprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Active Comparator): hrIL-2 active (1 million U doses of hrIL-2s.c.injection) MTX Folic acid Loxoprofen
  Interventions: Drug: hrIL-2 active; Drug: MTX; Drug: Folic Acid; Drug: Loxoprofen
- Placebo Comparator (Placebo Comparator): hrIL-2 placebo (1 million U doses of placebo s.c.injection) MTX Folic acid Loxoprofen
  Interventions: Drug: hrIL-2 placebo; Drug: MTX; Drug: Folic Acid; Drug: Loxoprofen

INTERVENTIONS:
Drug: hrIL-2 active — hrIL-2 active (1 million U doses of hrIL-2s.c.injection)
  Other Names: Human recombinant IL-2
  Arms: Experimental
Drug: hrIL-2 placebo — hrIL-2 placebo (1 million U doses of hrIL-2 placebo s.c.injection)
  Other Names: placebo
  Arms: Placebo Comparator
Drug: MTX — Methotrexate (oral administration)
Drug: Folic Acid — Folic Acid (oral administration)
Drug: Loxoprofen — Loxoprofen (oral administration)

SUMMARY:
Rheumatoid arthritis (RA) is an immune-mediated inflammatory disease, characterized by symmetric poly-arthritis usually involving the small joints of the hands and feet. In addition, various extra-joint manifestations may develop. Several immunomodulating agents have been attempted in the treatment of RA without achieving satisfactory results. Dysfunction of regulatory T (Treg) cells has been detected in diverse autoimmune diseases, which can be promoted by interleukin-2 (IL-2). The investigators hypothesized that low-dose IL-2 could be a novel therapy in active RA patients. This clinical study will test the efficacy and safety of low dose IL-2 treatment in RA. The investigators perform a single-centre, double-blind pilot trial with hrIL-2 in RA. The investigators evaluate the effectiveness and safeness of low-dose hrIL-2 for RA by randomized controlled study (hrIL-2 (N = 23) + Methotrexate (MTX)+ Loxoprofen versus placebo+MTX + Loxoprofen group (N = 24)).

DETAILED DESCRIPTION:
Each RA patients (n=47) with DAS>3.2 received low-dose IL-2+MTX+ Loxoprofen or placebo+MTX + Loxoprofen (active group: placebo group =1:1, 1 million units every other day subcutaneously (hrIL-2 1×106, ip, Qod) for a period of 14 days. After a 14-day rest, another cycle started) for 3 cycles. The end points were safety and clinical and immunologic response.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 and ≤70 years of age at time of screening
* Diagnosed with rheumatoid arthritis
* Must have active disease with DMARDs (Disease Modifying Anti-Rheumatic Drugs) except MTX, the doses had been stable for at least 3 months before baseline
* Moderate or severe rheumatoid arthritis during screening, as defined by a disease activity score (28 joint) calculated using the C-reactive protein formula (DAS28-ESR) > 3.2
* Have given written informed consent

Exclusion Criteria:

* Patient presenting or having a history of other inflammatory joint disease
* Patient with ongoing or previous Stevens-Johnson syndrome, toxic epidermal necrolysis or erythema multiforme
* Patient with significantly impaired bone marrow function or significant anaemia, leucopenia or thrombocytopenia due to causes or other than active rheumatoid arthritis
* Persistent infection or severe infection within 3 months before enrollment,
* Uncontrolled hypertension, uncontrolled diabetes, unstable ischemic heart disease, active inflammatory bowel disease, active peptic ulcer disease, terminal illness or other medical condition which, in the opinion of the investigator, would put the patient at risk to participate in the study,
* Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult
* Severe hypoproteinemia (e.g., in case of severe liver disease or nephrotic syndrome) with serum albumin < 30 g/L
* Moderate or severe impairment of renal function, as known by serum creatinine > 133μmol/L (or 1.5 mg/dl)
* Patient with history of recent and clinically significant drug or alcohol abuse
* Impairment of liver function or persisting ALT (SGPT) elevations of more than 2-fold the upper limit of normal
* Known HIV positive status
* Known positive serology for hepatitis B or C
* Patient with hypersensitivity to any of the excipients in the tablets of methotrexate
* Pregnancy
* Breastfeeding
* Women of childbearing potential, except if they fulfill specific conditions,
* Men wishing to father children during the course of the study or within the 24 months thereafter (or 3 month with the washout procedure)
* Patient with a congenital or acquired severe immuno-deficiency, a history of cancer or lymphoproliferative disease, or any patient who has received total lymphoid irradiation.
* Enrollment in any other clinical trial involving off-label use of an investigational drug or device, or enrollment in any other type of medical research
* Any active infection (including chronic or localized infections) for which anti-infectives were indicated within 28 days prior to first investigational product dose
* BMI(body mass index) under 18.5 kg/m2 or more than 30 kg/m2
* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, MD PhD, Principal Investigator — Peking University Institute of Rheuamotology and Immunology
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang X, Miao M, Zhang R, Liu X, Zhao X, Shao M, Liu T, Jin Y, Chen J, Liu H, Zhang X, Li Y, Zhou Y, Yang Y, Li R, Yao H, Liu Y, Li C, Li Y, Ren L, Su Y, Sun X, He J, Li Z. Efficacy and safety of low-dose interleukin-2 in combination with methotrexate in patients with active rheumatoid arthritis: a randomized, double-blind, placebo-controlled phase 2 trial. Signal Transduct Target Ther. 2022 Mar 7;7(1):67. doi: 10.1038/s41392-022-00887-2. PMID 35250032

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental | Placebo Comparator
Started | 23 | 24
Completed | 17 | 23
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Placebo Comparator | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (10.9) | 56.4 (9.9) | 54.5 (10.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 20 | 20 | 40
  Sex: Male | 3 | 4 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving DAS28 Remission.
Description: DAS 28 remission is defined by a disease activity score (28 joint) calculated using the erythrocyte sedimentation rate (DAS28-ESR) of less than 2.6
Time Frame: week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
Participants | 6 | 6
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.530, Chi-squared

2. Primary Outcome: Percentage of Participants Meeting the American College of Rheumatology 20% Response Criteria
Description: The assessments are based on a 20% or greater improvement from Baseline in the number of tender joints, a 20%, or more improvement in the number of swollen joints, and a 20% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: week 12, week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
Participants
  week 24 | 13 | 13
  week 12 | 12 | 10
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.315, Chi-squared

3. Primary Outcome: The Change From Baseline of Clinical Disease Activity Index (CDAI)
Description: Clinical Disease Activity Index(CDAI), the minimum is 0, the maximum is 76. higher scores mean a worse outcome.
  The change of from baseline of CDAI, the minimum is -76, the maximum is 76. higher scores mean a worse outcome.
Time Frame: week 12, week 24
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
score on a scale
  week 24 | -17.5 [-22 to -11] | -11 [-17.5 to -7.0]
  week 12 | -15.0 [-19.0 to -9.7] | -8.0 [-16.9 to -3.5]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.018, Mixed Models Analysis

4. Primary Outcome: The Change From Baseline of Simplified Disease Activity Index (SDAI)
Description: Simplified Disease Activity Index(SDAI). the minimum is 0, the maximum is 96. higher scores mean worse outcome.
  The change from baseline of SDAI. the minimum is -96, the maximum is 96. higher scores mean worse outcome.
Time Frame: week 12, week 24
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
score on a scale
  week 24 | -19.0 [-23.1 to -12.2] | -12.1 [-19.3 to -6.3]
  week 12 | -16.9 [-19.1 to -9.8] | -9.2 [-17.2 to -3.9]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.015, Mixed Models Analysis

5. Secondary Outcome: Number of Participants With Adverse Events
Description: adverse events includes injection site reactions, influenza-like symptoms, infection, fever, tumor, cardiovascular event, drug-induced liver and kidney damage.
Time Frame: Up to week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 23 | 24
Participants | 11 | 9
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other — Chi; p = 0.474, Chi-squared

6. Secondary Outcome: Percentage of CD4+ Treg Cells
Description: analysis regulatory CD4+ T(Treg) cells before and during IL-2 treatment. P values<0.05 are considered statistically significant.
Time Frame: week 12, week 24
Measure: Mean (Full Range); unit: percentage of CD4+ T cells
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
percentage of CD4+ T cells
  Week 24 | 6.94 [2.18 to 13.77] | 6.46 [3.71 to 12.30]
  Week 12 | 6.84 [3.7 to 10.61] | 5.37 [3.2 to 7.86]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other — description of Treg cells in CD4+ T cells; p = 0.665, Mixed Models Analysis

7. Secondary Outcome: Percentage of Participants Achieving DAS28 Low Disease Activity.
Description: Low disease activity is defined by a disease activity score (28 joint) calculated using the erythrocyte sedimentation rate (DAS28-ESR) of less than 3.2
Time Frame: week 12, week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
Participants
  week 24 | 8 | 9
  week 12 | 7 | 7
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.616, Chi-squared

8. Secondary Outcome: Percentage of Participants Achieving a Good or Moderate European League Against Rheumatism (EULAR) Response
Description: Good response is defined as: DAS28-ESR ≤ 3.2 and decrease from Baseline by > 1.2.
  moderate response is defined as achievement of one of the following: DAS28-ESR ≤ 3.2 and decrease from Baseline > 0.6 and ≤ 1.2 DAS28-ESR > 3.2 and ≤ 5.1 and decrease from Baseline > 0.6 DAS28-ESR > 5.1 and decrease from Baseline >1.2.
Time Frame: week 12, week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
Participants
  week 24 | 17 | 20
  week 12 | 15 | 14
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.616, Chi-squared

9. Secondary Outcome: Percentage of Participants Meeting the American College of Rheumatology 50% Response Criteria
Description: The assessments are based on a 50% or greater improvement from Baseline in the number of tender joints, a 50%, or more improvement in the number of swollen joints, and a 50% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: week 12, week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
Participants
  week 24 | 10 | 8
  weed 12 | 6 | 3
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.200, Chi-squared

10. Secondary Outcome: Percentage of Participants Meeting the American College of Rheumatology 70% Response Criteria
Description: The assessments are based on a 70% or greater improvement from Baseline in the number of tender joints, a 70%, or more improvement in the number of swollen joints, and a 70% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: week 12, week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
Participants
  week 24 | 4 | 2
  week 12 | 2 | 0
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.373, Chi-squared

11. Secondary Outcome: Percentage of Participants Meeting the 2011 American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) Remission Criteria Simplified for Clinical Practice
Description: The 2011 ACR/EULAR remission criteria simplified for clinical practice is defined as:Tender Joint Count (TJC) ≤ 1, Swollen Joint Count (SJC) ≤ 1 and Patient's Global Assessment of Disease Activity (PtGADA) ≤ 1.
Time Frame: week 12, week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
Participants
  week 24 | 2 | 1
  week 12 | 0 | 0
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.565, Chi-squared

12. Secondary Outcome: The Change From Baseline of a Health Assessment Questionnaire- Disability Index (HAQ-DI)
Description: The domains of the HAQ-DI are dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. The total score ranges from 0 to 3 with lower scores meaning lower disability.
  The change from baseline of HAQ-DI, minimum is -3, the maximum is 3. higher scores mean a worse outcome.
Time Frame: week 12, week 24
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
score on a scale
  week 24 | -0.63 [-0.88 to -0.13] | -0.38 [-0.75 to 0]
  week 12 | -0.50 [-0.88 to -0.19] | -0.25 [-0.63 to 0.00]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.221, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: The Scores of SF-36 Quetionnaire
Description: Score ranging from 0 to 100 with higher scores a better outcome.
Time Frame: week 12, week 24
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
score on a scale
  week 24 | 15.29 [8.73 to 29.65] | 6.90 [1.39 to 16.61]
  week 12 | 24.32 [11.89 to 40.85] | 27.25 [16.58 to 41.47]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.085, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]
Description: The Arthritis interference in the last month with work productivity is measured on a scale that ranges from 0 (no interference) to 10 (complete interference). The Arthritis interference in the last month with household work productivity is measured on a scale that ranges from 0 (no interference) to 10 (complete interference).higher scores mean a worse outcome.
Time Frame: week 24
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 23 | 24
units on a scale
  rate of Arthritis interference | 3 [0 to 6.75] | 2 [0 to 6.5]
  Rate of arthritis interference with household work | 5 [3 to 10] | 5 [2.25 to 6]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.740, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Time Frame: week 12, week 24
Measure: Mean (Standard Deviation); unit: millimeter/hour
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
millimeter/hour
  Week 24 | 43.3 (25.9) | 36.8 (24.9)
  Week 12 | 29.6 (25.6) | 28.3 (21.6)
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.881, Mixed Models Analysis

16. Secondary Outcome: C Reactive Protein (CRP)
Time Frame: week 12, week 24
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
mg/L
  week 24 | 21.6 (20.83) | 15.32 (14.74)
  week 12 | 9.5 (9.0) | 7.8 (7.2)
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.422, Mixed Models Analysis

17. Secondary Outcome: The Change From Baseline of Patient's Global Assessment of Disease Activity (PtGADA)
Description: VAS score from 0 to 100 for Patient's Global Assessment of Disease Activity Higher scores mean a worse outcome. The change from baseline of PtGADA, the minimum is -100, the maximum is 100. Higher scores mean a worse outcome.
Time Frame: week 12, week 24
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
score on a scale
  week 24 | -57.5 [-76.4 to -29.5] | -33.3 [-66.7 to 0]
  week 12 | -57.1 [-75.0 to -35.4] | -33.3 [-62.5 to 0.0]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.055, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: The Change From Baseline of Physician's Global Assessment of Disease Activity (PhGADA)
Description: VAS score from 0 to 100 for Physician's Global Assessment of Disease Activity higher scores mean a worse outcome. The change from baseline, the minimum is -100, the maximum is 100.
Time Frame: week 12, week 24
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
score on a scale
  week 24 | -58.3 [-76.4 to -47.2] | -44.4 [-57.1 to 0.0]
  week 12 | -57.1 [-66.7 to -33.3] | -25.0 [-44.4 to 0.0]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.039, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: The Change From Baseline of Patient's Assessment of Arthritis Pain (PtAAP)
Description: VAS score from 0 to 100 for Patient's Assessment of Arthritis Pain higher scores mean a worse outcome. The change from baseline of PtAAP, the minimum is -100, the maximum is 100.
Time Frame: week 12, week 24
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 17 | 23
score on a scale
  week 24 | -57.5 [-76.4 to -29.5] | -33.3 [-66.7 to 0.0]
  week 12 | -57.1 [-69.6 to -41.5] | -27.3 [-42.7 to 0.0]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Other; p = 0.156, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]-2
Description: In the last month, number of work days missed, number of work days with reduced productivity. In the last month, number of days with no household work, number of days with reduced household work productivity, number of days with hired outside help, number of days missed of family/social/leisure activities in the last month.higher scores mean a worse outcome.
Time Frame: week 24
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 23 | 24
days
  number of work days with reduced productivity | 3.5 [0 to 20] | 0 [0 to 18]
  number of work days missed | 0 [0 to 0] | 0 [0 to 0]
  Household work days missed due to arthritis | 0 [0 to 10] | 0 [0 to 6.5]
  Days with household work productivity reduced | 15 [3 to 30] | 12 [5 to 30]
  Days with activities missed due to arthritis | 5 [0 to 7] | 0 [0 to 7]
  Days with outside help hired due to arthritis | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Arm/Group | Experimental | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 11/23 | 9/24
Serious Adverse Events (participants affected / at risk) | 2/23 | 1/24
Other Adverse Events (participants affected / at risk) | 9/23 | 8/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=23) | Placebo Comparator (N=24)
Hospitalized not related to RA (Surgical and medical procedures) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=23) | Placebo Comparator (N=24)
gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hepatic enzyme increased (Hepatobiliary disorders) | 1 (1) | 1 (1)
Injection site reactions (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Fever after injection (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Worsening of RA (Immune system disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes